CLINICAL TRIAL: NCT03935412
Title: The Analgesic Efficacy of Bilateral Erector Spinae Plane Block in Comparison With Intrathecal Morphine After Elective Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Mohamed hamed, mohamed ahmed hamed, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R 125
Record Dates: First submitted 2019-03-01; First posted 2019-05-02 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Postoperative Pain
Keywords: Erector spinae plane block; morphine; cesarean section; postoperative analgesia; spinal anesthesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ES Erector Spinae Plane Block (Active Comparator): By the end of surgery parturient in the ESPB underwent bilateral ESPB at the level of T9 using a linear ultrasound (US) transducer (Phillips Saronno Italy) the transducer was placed vertically3cm lateral to the midline to visualize the muscles of the back, transverse process and the pleura in between the two transverse processes. After local infiltration of the needle insertion site with 2-3 ml of 2% lidocaine 22-G short bevel needle (spinocan, B.Braun melsungen AG, Germany) was inserted in cranial-caudal direction towards the transvers process using in plane technique until the needle cross all the muscles then interfascial injection of 20ml 0.5% bupivacaine was done after ensuring negative aspiration, the procedure was repeated following the same steps on the other side of the back.
  Interventions: Procedure: Erector Spinae Plane Block
- intrathecal morphine ITM (Sham Comparator): participant in the ITM group intrathecal injection of 10mg of hyperbaric bupivacaine 0.5 % in addition to 100 mcg of preservative-free morphine. Then, the parturient immediately placed in the supine position with 15° left tilt, and an oxygen mask was applied at 2 l.min-1. After ensuring sufficient anesthesia level, the surgical procedure was done with continuous hemodynamics monitoring and recording. While participants in the ITM group underwent sham blocks; Sham blocks consisted of a non-invasive ultrasound scan, while a blunt needle was gently pressed on both sides.
  Interventions: Procedure: Erector Spinae Plane Block

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — Erector Spinae Plane Block

SUMMARY:
The aim of this study was to assess the analgesic efficacy of bilateral erector spinae plane block in comparison with intrathecal morphine after elective cesarean section under spinal anesthesia.

DETAILED DESCRIPTION:
140 parturient scheduled for elective cesarean section. We obtained a written informed consent for anesthesia from each patient after explaining to them the nature of study and possible complications. Parturient were eligible for enrollment if they met the following inclusion criteria: Parturient aged 18 - 40 years , with American Society of Anesthesiologists physical status (ASA) class Ι, scheduled for elective cesarean section via a low transverse abdominal incision (Pfannenstiel) and receiving intrathecal anesthesia without sedation. Exclusion criteria included significant hepatic, renal or cardiovascular diseases, local infection, bleeding disorders, any contraindication to intrathecal anesthesia and parturient had a known allergy to the study drugs.

Participants were randomly divided into two groups (ITM; intrathecal morphine and ESPB; erector spinae plane block groups, with 70 participants in each) as simple randomization by computer-generated random numbers that were placed in separate opaque envelopes opened by responsible anesthesiologist just before intrathecal block. The participants, the study investigators and the data collectors were not aware of group allocation till the study end. Those in the ITM group were given 100 mcg of preservative-free morphine in addition local anesthetic (hyperbaric bupivacaine 10 mg) intrathecally during spinal anesthesia. While participants in the ESPB group were given only local anesthetic (hyperbaric bupivacaine 10 mg) intrathecally.

Preoperative investigations including electrocardiogram (ECG), complete blood picture, renal function tests, liver function tests, and coagulation profile were done. All parturient were fast for 8 h preoperatively. Upon arrival to the operating room IV access was obtained (one peripheral venous cannula 18G) and standard monitoring including pulse oximetry, ECG and noninvasive blood pressure were placed. And 10 ml.kg-1 of Ringer lactate solution will be infused over 15 minutes as a preload. The responsible anesthesiologist then asked the parturient to turn into sitting position where the skin on the back sterilized and; Spinal anesthesia performed via a midline approach into the L4-5 interspaces using a 25 gauge Quincke spinal needle after giving 3 ml of lidocaine 2% as a subcutaneous infiltration. After confirming free CSF flow through the needle a 10mg of hyperbaric bupivacaine 0.5 % was slowly injected for those in the ESPB group; and for those in the ITM group intrathecal injection of 10mg of hyperbaric bupivacaine 0.5 % in addition to 100 mcg of preservative-free morphine. Then, the parturient immediately placed in the supine position with 15° left tilt, and an oxygen mask was applied at 2 l.min-1. After ensuring sufficient anesthesia level, the surgical procedure was done with continuous hemodynamics monitoring and recording. If the systolic blood pressure (SBP) decreased to 20% below the baseline or less than 90 mmHg, ephedrine 5 mg will be administered intravenously. Also, if HR will be less than 50 beats/ min, atropine sulfate 0.5 mg will be administered intravenously. Upon delivery of the fetus, ten units of oxytocin were given by IV infusion.

By the end of surgery parturient in the ESPB underwent bilateral ESPB at the level of T9 using a linear ultrasound (US) transducer (Phillips Saronno Italy) the transducer was placed vertically3cm lateral to the midline to visualize the muscles of the back, transverse process and the pleura in between the two transverse processes. After local infiltration of the needle insertion site with 2-3 ml of 2% lidocaine 22-G short bevel needle (spinocan, B.Braun melsungen AG, Germany) was inserted in cranial-caudal direction towards the transvers process using in plane technique until the needle cross all the muscles then interfascial injection of 20ml 0.5% bupivacaine was done after ensuring negative aspiration, the procedure was repeated following the same steps on the other side of the back. While participants in the ITM group underwent sham blocks; Sham blocks consisted of a non-invasive ultrasound scan, while a blunt needle was gently pressed on both sides. We instructed the participants to report any signs of local anesthetic toxicity throughout injection e.g. change in mental status, anxiety, oral numbness and ringing in ears. For all participants spinal level and numerical rating scale were assessed and recorded before the block. At the end of surgery, parturient were transferred to postoperative anesthesia care unit (PACU) with standard monitoring applied. Any intraoperative or postoperative nausea or vomiting was managed with 10 mg metoclopramide. All participants received 30 mg ketorolac intravenously with the time of ESPB or sham blocks. Participants were transferred to obstetrics ward after fulfilling the criteria of modified Aldrete scoring system.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status (ASA) class Ι, scheduled for elective cesarean section via a low transverse abdominal incision (Pfannenstiel) and receiving intrathecal anesthesia without sedation

Exclusion Criteria:

* included significant hepatic, renal or cardiovascular diseases, local infection, bleeding disorders, any contraindication to intrathecal anesthesia and parturient had a known allergy to the study drugs.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-05 (Actual)

PRIMARY OUTCOMES:
the severity of pain: VAS | 8 hour
  VAS

SECONDARY OUTCOMES:
the total analgesic consumption | 24 hour
  AMOUNT
the severity of pain: VAS | immediately in PACU
  VAS
the severity of pain: VAS | 4 hours
  VAS
the severity of pain: VAS | 12 hours
  VAS
the severity of pain: VAS | 16 hours
  VAS
the severity of pain: VAS | 24 hours
  VAS
the time for the first analgesic request | 24 hours
  time
Participants' satisfaction | 24 hours
  postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Al Fayyum, Egypt

REFERENCES:
- [Background] Ueshima H, Otake H. Similarities Between the Retrolaminar and Erector Spinae Plane Blocks. Reg Anesth Pain Med. 2017 Jan/Feb;42(1):123-124. doi: 10.1097/AAP.0000000000000526. No abstract available. PMID 27997492
- [Result] Leung AY. Postoperative pain management in obstetric anesthesia--new challenges and solutions. J Clin Anesth. 2004 Feb;16(1):57-65. doi: 10.1016/j.jclinane.2003.02.012. PMID 14984863